CLINICAL TRIAL: NCT07174869
Title: A Pilot Study To Assess The Dynamic Difficulty Adjustment In Personalized Testing For Persons With MCI And Matched Healthy Controls
Brief Title: A Study To Assess The Feasibility Of Indivi Mobile Application In Monitoring Cognitive Performance In Aging Population
Acronym: ADAPT-MCI-01
Status: Recruiting | Type: Observational
Sponsor: Indivi AG (Industry)
Responsible Party: Sponsor
Other Study IDs: H-45373
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment (MCI); Mild Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PwMCI/AD: Persons with Mild Cognitive Impairment or mild Alzheimer's Disease
- HC: Healthy Controls

SUMMARY:
The goal of this observational study is to evaluate the functionality and usability of Indivi mobile application-based cognitive activities in people with mild cognitive impairment/mild Alzheimer's disease (PwMCI/AD) and healthy controls (HC). This application uses a dynamic difficulty adjustment (DDA) system that customizes the level of the cognitive activities to each user.

The main questions it aims to answer are:

* Does the DDA system reach a stable difficulty level at the same rate for both PwMCI/AD and HC?
* Is the stable difficulty level reached by the DDA system different for PwMCI/AD compared to HC?

Researchers will also compare cognitive activities results and other aspects of the mobile application's performance to see if the application can validly distinguish between the two groups.

Participants will use the Indivi mobile application, with its embedded DDA system, for a 6-week period.

ELIGIBILITY:
Inclusion Criteria:

* Participant is part of BU-ADRC cohort.
* Participant is diagnosed with MCI, mild AD, or is classified as HC per BU-ADRC, with available required data for inclusion obtained less than 2 years before the inclusion.
* Participant is between 50 and 90 years old, included.
* Participant is able to use a smartphone.
* Participant has sufficient knowledge of the English language.
* Participant is able to and has an intention to follow the study procedures.
* Informed Consent as documented by signature.

Exclusion Criteria:

* Participant has any neurological condition that may be contributing to cognitive impairment (above and beyond that caused by the subject's MCI or AD).
* Participant has psychiatric diagnosis or symptoms, (e.g., hallucinations, major depression, or delusions) that could interfere with study procedures.
* Participant has a history of stroke or seizures within the last 24 months.
* Participant has a Geriatric Depression Scale (GDS) score ≥8.
* Participant has a severe visual or hearing impairment that would interfere with capacity to perform cognitive assessments.
* Known or suspected non-compliance.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Boston University Alzheimer's Disease Research Center (BU ADRC)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of test iterations until stable difficulty level is reached | During the 6-week study period.
  Stable difficulty level is defined as no increase in difficulty across 3 consecutive test iterations. Comparison will be made between PwMCI and HC.
Distribution of participants across assessment levels at steady-state difficulty | During the 6-week study period
  Steady-state difficulty is defined as no increase in difficulty across 3 consecutive test iterations. The outcome will describe the distribution pattern of participants across the available assessment levels at steady-state.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes